CLINICAL TRIAL: NCT01589445
Title: Modulation of Insulin Secretion and Insulin Sensitivity in Bangladeshi Type 2 Diabetic Subjects by an Insulin Sensitizer Pioglitazone and T2DM Association With PPARG Gene Polymorphism.
Brief Title: Efficacy Study of Pioglitazone and Metformin and Association Between Pioglitazone Response and Peroxisome Proliferator-activated Receptor Gamma Gene Variants in Bangladeshi Type 2 Diabetes Mellitus Subjects
Acronym: T2DMCT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Dhaka (Other)
Collaborators: Bangladesh Institute of Research and Rehabilitation in Diabetes, Endocrine and Metabolic Disorders (Other); University of Dundee (Other)
Responsible Party: Principal Investigator, Dr. Masuma Parvin, Research fellow, University of Dhaka
Allocation: Non-Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BS-67/2008-09; BMRC/ERC/2007-2010/2024 (Other: Bangladesh Medical Research Council)
Record Dates: First submitted 2012-04-29; First posted 2012-05-02 (Estimated); Results first posted 2014-02-27 (Estimated); Last update posted 2014-02-28 (Estimated); Status verified 2014-02

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Bangladesh; T2DM; Pioglitazone; Metformin; Insulin secretion and Sensitivity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypersensitivity | interventions — Pioglitazone; Tablets; Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pioglitazone (001 group) (Experimental): The patients received pioglitazone hydrochloride tablet 30 mg (001 drug)once daily for first three months
  Interventions: Drug: Pioglitazone hydrochloride; Drug: Metformin hydrochloride
- Metformin (002 group) (Experimental): The patients received metformin hydrochloride tablet 850 mg (002 drug)once daily for next three months.
  Interventions: Drug: Pioglitazone hydrochloride; Drug: Metformin hydrochloride

INTERVENTIONS:
Drug: Pioglitazone hydrochloride — 77 patients were treated with pioglitazone hydrochloride (B001) for 3 months.Biomedical parameters were measured each month.
  Other Names: GLUCOZON; 30 mg tablet, once, daily; Coded as B001(Preparation Date:Jun 08); Aristopharma LTD.,Bangladesh
Drug: Metformin hydrochloride — After the treatment with pioglitazone(001) for 3 months first and then patients were on one month washout period;in the washout period they were given metformin tablet 850mg once daily,then treated with 002 (metformin) for further 3 months. The same biomedical measurements were assayed.
  Other Names: GLUCOMET; 850 mg tablet, once, daily; Coded as B002 (Preparation date: Jun 08); Aristopharma LTD.,Bangladesh

SUMMARY:
* The present study was undertaken to assess the efficacy and safety of two different insulin sensitizers (namely Pioglitazone and Metformin) among subjects with type 2 diabetes mellitus (T2DM) in Bangladesh.
* A prospective, double-blind, single group, 'within-subject' designed clinical trial of 77 diagnosed T2DM patients out of 130 patients with glycosylated haemoglobin (HbA1c) ≥7.2±1.5%, aged 46±6.4 years and registered for diabetes treatment in Bangladesh Institute of Research and Rehabilitation in Diabetes Endocrine and Metabolic Disorders (BIRDEM) was carried out.
* The study was conducted between November 2008 and September 2010.
* Baseline data, included case history of the patients,anthropometric measurement, biomedical parameters psychosocial factors, were collected from each subject and then enrolled to receive treatment with 001 drug once daily for three months, then the patients were left for wash out with metformin 850mg once daily for one month; then they received 002 drug once daily for further three months.
* Dietary chart was remained as before.
* DNA was isolated by Chelex method using the primers and control DNA,restriction Digestion Enzyme Endonuclease Hae 111 for genotyping PPARγ-(Peroxisome Proliferator Activated Receptor gamma)Pro12Pro

  * (Proline12Proline)/Pro12Ala-(Proline12 Alanine))/Ala12Ala-(Alanine12Alanine).
* The blinded drugs were decoded after analyzing results, 001 tablet was pioglitazone (30 mg once daily) and 002 tablets was metformin (850mg once daily). Bio-medical outcomes were measured to assess the efficacy of both the drugs each month. After finishing the treatment period the effects of two drugs were compared using SPSS.And the association between the pioglitazone drug effects and genetic polymorphism was also assessed.
* The metformin effects was assessed also using the response rate of HbA1c <7.0% after 3 months treatment to the patients.

DETAILED DESCRIPTION:
1. Introduction Thiazolidinediones and metformin are known drugs and especially metformin is widely used medicine to treat people with T2DM. Though pioglitazone has been suspended in many countries, its safety and efficacy is a matter of research for the drug investigators. Thiazolidinediones had been introduced in 1997 as an oral anti-diabetic drug (OAD). Metformin has been used as the key compound to treat T2DM for many years and is the most prescribed OAD worldwide. Both metformin and thiazolidinediones are considered as "insulin sensitizer". The ß-cell dysfunction and insulin resistance are the core defects in the progression of T2DM with associated metabolic syndrome. Evidence suggests that pioglitazone lowers glucose in blood by increasing glucose uptake into cell and metformin by decreasing glucose production. However, there are many controversies in clinical study specially about the improvement of insulin action of metformin. In contrast, a research recommended pioglitazone as the most appropriate OAD for the South Asian population. The key to this argument is that since pioglitazone is a proliferator-activated receptor gamma (PPAR-γ or PPARG) [a group of nuclear receptor proteins that function as transcription factors regulating the expression of genes] agonist and decreases insulin resistance, overall glycemic control seems to be better with this thiazolidinedione. However, there are very few published documents on the efficacy and safety of these drugs in South Asians. To the best of our knowledge, there is no published paper that examined and compared the efficacy and safety of these two drugs in Bangladeshi patients T2DM. This double-blind trail therefore examined the efficacy and safety of pioglitazone and metformin in T2DM individuals and also the association of the effects of pioglitazone and the variants of PPARG. We have compared the effects of pioglitazone with metformin on biomedical variables in T2DM patients who were eligible for oral hypoglycaemic therapy and then we also analyzed the association among the effects of pioglitazone and PPARG variants.
2. Methodology

   1. Study Setting:

      The study was conducted between November 2008 and September 2010. The participants for this study were recruited from the outdoor, BIRDEM Hospital in Dhaka,Bangladesh.
   2. Subjects I.Individuals who had been diagnosed with T2DM treating with diet/exercise or Metformin 850 mg or Pioglitazone 30mg once daily, and were attending Outdoor Patient Department (OPD) of BIRDEM for consultation were approached by the researcher and invited to participate in the study. The patients were diagnosed already and registered in BIRDEM. T2DM was ascertained based on World Health Organization recommended criteria two repeated measures of fasting (plasma glucose ≥7.0 mmol ⁄ l or 2-h plasma glucose ≥11.1 mmol ⁄ l.)

      II.We screened a total of 130 patients for eligibility and selected 80 patients for enrollment based of our inclusion and exclusion criteria. But 77 T2DM patients with HbA1c level < 7.5 %, BMI kg/m2 ≥ 25, SGPT≤ 100 IU/L , creatinine ≤ 1.2 mg/dl) of both sexes, aged between 40-50, treated by monotherapy of pioglitazone or metformin received the drug for the trial according to inclusion and exclusion criteria. 53 patients were screening failure as some did not match eligibility criteria (n=39), some refused to take part(n=11)and some were unable to take part (n=03)due to unknown cause.
   3. Patient Preparation:

      I.Written informed consent was obtained from all participants before study entry. Patients were instructed to follow adhere to a disease- and weight-orientated diet throughout the study as before.

      II.Each case history was documented in the case report form. The study was approved by the National Medical Ethics Review Boards (NMERB) of Bangladesh Medical Research Council (BMRC).The investigations were carried out in accordance with the principles of the Declaration of Helsinki as revised in 2000.
   4. Treatment:

      The patients were to receive treatment pioglitazone tablet 001 (30mg once per day) for 3 months followed by one month "metformin wash-out period", then to the alternative treatment regimen for further 3 months with metformin tablet 002 (850mg once per day). The drugs were supplied by the Aristopharma Pharmaceutical Ltd., Bangladesh.
   5. Anthropometric Measurements I.Height: Standing height was measured using appropriate scales (Detect-Medic, Detect scales INC, USA) without shoes.

      II.Weight: Weight was measured with the balance was placed on a hard flat surface and checked for zero balance before measurement. The subjects were in the center of the platform wearing light cloths without shoes.

      III.BMI: Body mass indexes (BMI) of the subjects were calculated using standard formula: BMI= Weight (kg)/[Height (m)] 2.

      IV.Blood Pressure: Systemic and Diastolic pressure was measured according to WHO-IHS.
   6. Blood Sample Collection for Biochemical analysis :

      I. During the appointed date the patients came in the fasting condition. Fasting blood samples (10 ml) were drawn from the antecubital vein. The time was mentioned as 0 hour. Then the patients received drug. They were requested to swallow the tablet and have their breakfast according to their diet charts. Next blood sample had been drawn at 30 min and 2 hour and then they were provided the drugs for the whole month.

      II.The patients were requested to take the drug just before the breakfast every day for 29 days.

      III.From the fasting blood sample 1ml of blood was transferred in an EDTA containing tube for measurement of HbA1C and the rest of the blood was taken in an EDTA containing tube and centrifuged immediately.

      IV.Samples after processing were divided into two aliquots under sterile condition;one aliquot was sent for biochemical analysis for Fasting glucose, Lipid profile, Cholesterol, ALT, Insulin, Creatinine and another one was stored at -80 0C for further verification of results in case of any necessity.
   7. Biochemical Test Methods:

      I. Serum glucose (fasting, 1 and 2 hours) by Glucose Oxidase (GOD-PAP) method (Randox Laboratories Ltd., UK).

      II.Serum triglyceride by enzymatic colorimetric (GPO-PAP) method (Randox Laboratories Ltd., UK).

      III.Serum total cholesterol by enzymatic endpoint (Cholesterol Oxidase/ Peroxidase) method (Randox Laboratories Ltd., UK).

      IV.Serum HDL cholesterol by enzymatic colorimetric (Cholesterol CHOD-PAP) method (Randox Laboratories Ltd., UK) using micro-plate reader (Bio-Tec, ELISA).

      V.Serum creatinine by enzymatic colorimetric (GPO-PAP) method (Randox Laboratories Ltd., UK).

      VI.Serum alanine amino transferase (ALT) by UV method using ALT (GPT) opt.kit (Randox Laboratories Ltd., UK).

      VII.Serum insulin by enzyme linked immunosorbent assay (ELISA) method (Linco Research Inc., USA).

      VIII.Glycosylated Haemoglobin (HbA1c) by High Performance Liquid Chromatographic (HPLC) method.
   8. Blood sample collection for DNA analysis (PPARG gene):

   I.At the end of 3rd month of each treatment 1.5 ml of blood was taken in EDTA containing tube for genetic analysis and the whole blood specimen was collected in the vacuum collection tube containing EDTA, stored at -20 0C to - 80 0C.

   II.DNA was isolated by Chelex method, identified by electrophoresis method and amplified by using primers. We used a published document to select the primers for genotyping PPARγ Pro12Ala/Pro12Pro. The primers for the Pro12Ala SNP genotype, we amplified exon B using the reverse primer 5' CTG GAA GAC AAA CTA CAA GAG 3' and the forward primer 5' ACT CTG GGA GAT TCT CCT ATT GGC 3'. (Sigma product, Order No. SIGMA 03/11/09 4152936-F/185 PPARG-R 8006875247-1).

   III.Control DNA: Professor Colin Palmer Laboratory, Biomedical Research Institute ,University of Dundee Medical School, University of Dundee, Scotland, UK sent six control samples of 3 types control DNA genotyped for PPARG SNP rs 1801282 (Pro12Ala).

   IV.Restriction Digestion Enzyme Endonuclease Hae 111 was used to identify the cutting site(Sigma Product No. R 5628).
3. Response Rate:

1. The response rate was defined by the decrease of ≥10% FBG or by the decrease of ≥1% HbA1c from the baseline values.

ll.There was another response group was defined by the the HbA1c rate <7.0% after 3 months treatment with metformin only to find out the secondary failure rate of metformin.

4) Statistical Analysis: I.Statistical analysis was performed using SPSS (Statistical Package for Social Science) software for Windows version 18 (SPSS Inc, Chicago, Illinois, USA). Data were expressed as mean + SD (Standard Deviation).

II. Effects of drugs after 3 months treatment were analyzed using t pair tests. The groups were compared using one way ANOVA. If the p value was <0.05, the groups were compared using the student's t test for unpaired samples or χ2 test through univariate analysis for further verification. Correlation coefficient among the variables was tested using Pearson's test. Multivariate logistic regression analysis was performed to obtain the odds ratios and independent influencing factor for finding possible association between PPARγ genotypes and drug response in case of genetic analysis.

III.A p value <0.05 was considered significant for all tests. lv. The statistical analysis for within group study like PPARG response group and metformin secondary failure group has not been displayed here.

5) List of Abbreviations

AEs Adverse Events

ALT Alanine aminotransferase

BMI Body Mass Index

BMRC Bangladesh Medical Research Council

BIRDEM Bangladesh Institute of Research and Rehabilitation in Diabetes,Endocrine and Metabolic Disorder

BP Blood Pressure

DNA Deoxynucleic Acid

DBP Diastolic Blood Pressure

DM Diabetes Mellitus

EASD European Association for the Study of Diabetes

EDTA Ethylene Diamine Tetra Acetic acid

ELISA Enzyme Linked Immunosorbent Assay

FBG/FSG Fasting Blood Glucose/Fasting Serum Glucose

FSI Fasting Serum Insulin

2hBG 2 hours Blood Glucose

HbA1c Glycosylated Haemoglobin

HOMA percent B Homeostasis Model Assessment percentage of beta cell function HOMA percent S Homeostasis Model Assessment percentage of sensitivity

HOMA IR Homeostasis Model Assessment Insulin Resistance

HDL-C High Density Lipid Cholesterol

IU/L International Unit/Litre

LDL-C Low Density Lipid Cholesterol

ml millilitre

mm millimetre

mg/dl milligram/ decilitre

MLR Multiple Logistic Regression

OPD Outdoor Patient Department

OMIM Online Mendelian Inheritance in Man

OR Odds Ratio

PPARγ Peroxisome Proliferator Activated Receptor gamma

Pro12Pro Proline12Proline

Pro12Ala Proline 12 Alanine

Ala12Ala Alanine12Alanine

PCR Polymerase Chain Reaction

QUICKI Quantitative Insulin sensitivity Check Index

SD Standard Deviation

SPSS Statistical Package for Social Science

SBP Systolic Blood Pressure

TC Total Cholesterol

TG Triglyceride

T2DM Type 2 Diabetes Mellitus

TZD Thiazolidinedione

µl Microliter

WHO World Health Organization

ELIGIBILITY:
Inclusion Criteria:

* Type 2 DM patients (with HbA1c level < 8.5 %, BMI kg/m2 ≥ 25, SGPT ≤ 100 IU/L , creatinine ≤ 1.2 mg/dl) of both sexes,
* Aged between 40-50,
* Treated by monotherapy of pioglitazone or metformin.

Exclusion Criteria:

* Patients with diabetes secondary to another cause.
* Patients suffering from serious incurrent illness requiring systemic treatment.
* Patients suffering from any other infectious diseases.
* Patients with impaired kidney function (serum creatinine level more than 1.2mg/dl)
* Patients with impaired hepatic function (SGPT ≥ 100 IU/L).
* Patients with pulmonary insufficiency with hypoxaemia.
* Triglyceriadiamea (TG ≥ 150mg/dl).
* Bloodpressure > 180 mmHg (Systolic) or > 110 mmHg (diastolic).
* Positive history of drug or alcohol abuse.
* Pregnant women and willing to be pregnant shortly.

Ages: 40 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 77 (Actual)
Dates: Start 2008-11; Primary Completion 2009-12 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AK Azad Chowdhury, PhD, Study Chair — University of Dhaka, Bangladesh; Masuma Parvin, PhD, Principal Investigator — University of Dhaka, Bangladesh; Begum Rokeya, PhD, Study Director — BIRDEM,Dhaka,Bangladesh; Colin Palmer, PhD, Study Director — University of Dundee
Locations (1):
- Bangladesh Institute of Research and Rehabilitation in Diabetes, Endocrine and Metabolic Disorders (BIRDEM), Dhaka, Dhaka Division, Bangladesh

REFERENCES:
- [Background] Laakso M. Hyperglycemia and cardiovascular disease in type 2 diabetes. Diabetes. 1999 May;48(5):937-42. doi: 10.2337/diabetes.48.5.937. PMID 10331395
- [Background] Zimmet P, Alberti KG, Shaw J. Global and societal implications of the diabetes epidemic. Nature. 2001 Dec 13;414(6865):782-7. doi: 10.1038/414782a. PMID 11742409
- [Background] Wild S, Roglic G, Green A, Sicree R, King H. Global prevalence of diabetes: estimates for the year 2000 and projections for 2030. Diabetes Care. 2004 May;27(5):1047-53. doi: 10.2337/diacare.27.5.1047. PMID 15111519
- [Background] Trivedi B, Mazumdar JD, Bhatt, Hemavathi KG. Effect of Shilajit on blood glucose and lipid profile in alloxan-induced diabetic rats. Indian J Pharmacol 2004; 36: 373-376.
- [Background] Michael J, Fowler MD. Microvascular and Macrovascular Complications of Diabetes. Clinical Diabetes 2008; 26 : 77-82.
- [Background] Mahtab H, Khan AR, Latif ZA, Pathan F, Ahmed T. Guideline for care of Type 2 Diabetes Mellitus in Bangladesh. BIRDEM Clinical Research Group Publishing 2003.
- [Background] Silink M. The diabetes epidemic: The case for a resolution on diabetes. Diabetic Endocrine Journal 2006; 34:3-4.
- [Background] Krall LP. The wide world of diabetes. In: World book of diabetes in practice. Krall LP. (ed) v2 Amsterdam: Elsevier Science publishing; 1986.
- [Background] Diabetes Statistics -Diabetes help. http://www.diabetes.org.uk/Professionals/ Publications-reports-and-resources/Reports-statistics-and-case-studies/Reports/ Diabetes-prevalance-2010
- [Background] Shaw JE, Sicree RA, Zimmet PZ. Global estimates of the prevalence of diabetes for 2010 and 2030. Diabetes Res Clin Pract. 2010 Jan;87(1):4-14. doi: 10.1016/j.diabres.2009.10.007. Epub 2009 Nov 6. PMID 19896746
- [Background] American Diabetes Association (ADA). Diagnosis and Classification of Diabetes Mellitus. Diabetes Care 2005; 28: 37-42.
- [Background] Florez H. [Steps toward the primary prevention of type II diabetes mellitus. Various epidemiological considerations]. Invest Clin. 1997 Mar;38(1):39-52. Spanish. PMID 9235072
- [Background] Health Survey for England. http://www.heartstats.org/datapage.
- [Background] National Service Framework for Diabetes: Standards http:// www. technology adoptioncentre.nhs.uk/assets/_files/documents/mar_10/nhs__1268044698_Diabetes_NSF.pdf
- [Background] Abdella N, Al Arouj M, Al Nakhi A, Al Assoussi A, Moussa M. Non-insulin-dependent diabetes in Kuwait: prevalence rates and associated risk factors. Diabetes Res Clin Pract. 1998 Dec;42(3):187-96. doi: 10.1016/s0168-8227(98)00104-1. PMID 9925350
- [Background] Singh RB, Bajaj S, Niaz MA, Rastogi SS, Moshiri M. Prevalence of type 2 diabetes mellitus and risk of hypertension and coronary artery disease in rural and urban population with low rates of obesity. Int J Cardiol. 1998 Sep 1;66(1):65-72. doi: 10.1016/s0167-5273(98)00141-7. PMID 9781790
- [Background] Ramachandran A, Snehalatha C, Latha E, Manoharan M, Vijay V. Impacts of urbanisation on the lifestyle and on the prevalence of diabetes in native Asian Indian population. Diabetes Res Clin Pract. 1999 Jun;44(3):207-13. doi: 10.1016/s0168-8227(99)00024-8. PMID 10462144
- [Background] Pan XR, Li GW, Hu YH, Wang JX, Yang WY, An ZX, Hu ZX, Lin J, Xiao JZ, Cao HB, Liu PA, Jiang XG, Jiang YY, Wang JP, Zheng H, Zhang H, Bennett PH, Howard BV. Effects of diet and exercise in preventing NIDDM in people with impaired glucose tolerance. The Da Qing IGT and Diabetes Study. Diabetes Care. 1997 Apr;20(4):537-44. doi: 10.2337/diacare.20.4.537. PMID 9096977
- [Background] Ramachandran A, Snehalatha C, Mary S, Mukesh B, Bhaskar AD, Vijay V; Indian Diabetes Prevention Programme (IDPP). The Indian Diabetes Prevention Programme shows that lifestyle modification and metformin prevent type 2 diabetes in Asian Indian subjects with impaired glucose tolerance (IDPP-1). Diabetologia. 2006 Feb;49(2):289-97. doi: 10.1007/s00125-005-0097-z. Epub 2006 Jan 4. PMID 16391903
- [Background] McKeigue PM, Shah B, Marmot MG. Relation of central obesity and insulin resistance with high diabetes prevalence and cardiovascular risk in South Asians. Lancet. 1991 Feb 16;337(8738):382-6. doi: 10.1016/0140-6736(91)91164-p. PMID 1671422
- [Background] McKeigue PM, Miller GJ, Marmot MG. Coronary heart disease in south Asians overseas: a review. J Clin Epidemiol. 1989;42(7):597-609. doi: 10.1016/0895-4356(89)90002-4. PMID 2668448
- [Background] West KM, Kalbfleisch JM. Glucose tolerance, nutrition, and diabetes in Uruguay, Venezuela, Malaya, and East Pakistan. Diabetes. 1966 Jan;15(1):9-18. doi: 10.2337/diab.15.1.9. No abstract available. PMID 5907153
- [Background] Sayeed MA, Banu A, Haq JA, Khanam PA, Mahtab H, Azad Khan AK. Prevalence of hypertension in Bangladesh: effect of socioeconomic risk factor on difference between rural and urban community. Bangladesh Med Res Counc Bull. 2002 Apr;28(1):7-18. PMID 12587756
- [Background] Sayeed MA, Hussain MZ, Banu A, Rumi MA, Azad Khan AK. Prevalence of diabetes in a suburban population of Bangladesh. Diabetes Res Clin Pract. 1997 Jan;34(3):149-55. doi: 10.1016/s0168-8227(96)01337-x. PMID 9069566
- [Background] Abu Sayeed M, Banu A, Khan AR, Hussain MZ. Prevalence of diabetes and hypertension in a rural population of Bangladesh. Diabetes Care. 1995 Apr;18(4):555-8. doi: 10.2337/diacare.18.4.555. PMID 7497870
- [Background] Sayeed MA, Mahtab H, Khanam PA, Latif ZA, Banu A, Khan AK. Prevalence of diabetes and impaired fasting glucose in urban population of Bangladesh. Bangladesh Med Res Counc Bull. 2007 Apr;33(1):1-12. PMID 18246729
- [Background] Diabetic Association of Bangladesh. Statistical Year Book. July 2009-June 2010; p 250. web version is available at www.dab-bd.org.
- [Background] Gyas M. Interviewed by: Parvin M. 16 October 2011.
- [Background] Kahn SE, Porte DJ. The pathophysiology of type II (noninsulindependent) diabetes mellitus: implications for treatment. In: Porte D Jr, Sherwin RS editor(s). Ellenberg & Rifkin's Diabetes Mellitus. 5th ed. Stamford, Conneticut (U.S.A.): Appleton & Lange, 1997.
- [Background] Richter B, Bandeira-Echtler E, Bergerhoff K, Clar C, Ebrahim SH. Pioglitazone for type 2 diabetes mellitus. Cochrane Database Syst Rev. 2006 Oct 18;2006(4):CD006060. doi: 10.1002/14651858.CD006060.pub2. PMID 17054272
- [Background] DeFronzo RA. Lilly lecture 1987. The triumvirate: beta-cell, muscle, liver. A collusion responsible for NIDDM. Diabetes. 1988 Jun;37(6):667-87. doi: 10.2337/diab.37.6.667. No abstract available. PMID 3289989
- [Background] DeFronzo RA. Pathogenesis of type 2 diabetes: metabolic and molecular implication for identifying diabetes genes. In: American Diabetes Association, eds (Annual Review Of Diabetes), AlexandriaVA: American Diabetes 1998; 1-93.
- [Background] Kain K, Catto Aj. Trans-Cultural Medicine: Insulin Resistance Syndrome In South Asians. The British Journal of Diabetes & Vascular Disease 2002; 2: 398.
- [Background] WHO Expert Consultation. Appropriate body-mass index for Asian populations and its implications for policy and intervention strategies. Lancet. 2004 Jan 10;363(9403):157-63. doi: 10.1016/S0140-6736(03)15268-3. PMID 14726171
- [Background] Mathur SK, Rathore R, Chandra S, Sharma BB, Sharma L, Mathur P, Mathur M. Primary pioglitazone failure in Asian Indian diabetics is not related to common Pro12Ala polymorph of PPAR-gamma gene. Indian J Physiol Pharmacol. 2009 Apr-Jun;53(2):175-80. PMID 20112822
- [Background] Zinnat R. Role of Insulin Defficiency and Insulin Resistance in the Pathogenesis of Type 2 Diabetes in Young Bangladesh Subjects. M.Phil thesis. Bangladesh Institute of Research and Rehabilitation in Diabetes, Endocrine and Metabolic Disorders; 1999.
- [Background] Alhossainy K. (kalhossainy@gmail.com). As per our database. Parvin M (acmasuma@gmail.com) 21 July 2011.
- [Background] Thiazolidinedione http://en.wikipedia.org/wiki/Thiazolidinedione
- [Background] Bluher M, Lubben G, Paschke R. Analysis of the relationship between the Pro12Ala variant in the PPAR-gamma2 gene and the response rate to therapy with pioglitazone in patients with type 2 diabetes. Diabetes Care. 2003 Mar;26(3):825-31. doi: 10.2337/diacare.26.3.825. PMID 12610044
- [Background] Patlak M. New weapons to combat an ancient disease: treating diabetes. FASEB J. 2002 Dec;16(14):1853. No abstract available. PMID 12468446
- [Background] DeFronzo RA, Goodman AM. Efficacy of metformin in patients with non-insulin-dependent diabetes mellitus. The Multicenter Metformin Study Group. N Engl J Med. 1995 Aug 31;333(9):541-9. doi: 10.1056/NEJM199508313330902. PMID 7623902
- [Background] Goodman & Gilmans'. The Pharmacological basis of Therapeutics. 10th ed. International Edition, McGraw Hill; 2001: p1701, 1704, 1706.
- [Background] Lasker SP, McLachlan CS, Wang L, Ali SMK , Jelinek HF. Discovery, treatment and management of diabetes (Review Article). Journal of Diabetology Feb 2010; 1:1 http://www.journalofdiabetology.org/
- [Background] MacCracken J, Hoel D. From ants to analogues. Puzzles and promises in diabetes management. Postgrad Med. 1997 Apr;101(4):138-40, 143-5, 149-50. doi: 10.3810/pgm.1997.04.195. No abstract available. PMID 9126208
- [Background] Pickup JC, Willium G. The history of diabetes mellitus. In Textbook of diabetes. 3rd ed. Vol-1.Oxford London: Blackwell Science Limited; 2003.
- [Background] Kahn CR. Banting Lecture. Insulin action, diabetogenes, and the cause of type II diabetes. Diabetes. 1994 Aug;43(8):1066-84. doi: 10.2337/diab.43.8.1066. No abstract available. PMID 8039601
- [Background] Dabson M. Experiments and observations on the urine in diabetes. Med Obs Inq 1776; 5: 298-316.
- [Background] Barnett DM, Krall LP. The History of diabetes. In Joslin's diabetes Mellitus, 14th ed. Boston MA. Lipincott William and Wilkins; 2005.
- [Background] Stuart AR. Insulin and related medication. In Pharmacologic aspects of nursing. Paghiro, AM and Pagliaro, LA (eds). USA. The C.V. Mosby Company; 1988.
- [Background] Von Mering J, Minowski O. Diabetes mellitus nach pancreas extripation. Arch Exper Path Pharmacol Leipzig 1890; 26: 371-87.
- [Background] De Meyer J. Sur la signification physiologique de la secretion interne du pancreas. Zbl Physiol 1904;18:S826.
- [Background] Classification and diagnosis of diabetes mellitus and other categories of glucose intolerance. National Diabetes Data Group. Diabetes. 1979 Dec;28(12):1039-57. doi: 10.2337/diab.28.12.1039. No abstract available. PMID 510803
- [Background] World Health Organization. Definition, Diagnosis, Classification of Diabetes Mellitus and its Complications. Geneva: WHO 1999. Report of a WHO Consultation. Part1: Diagnosis and Classification of Diabetes Mellitus.
- [Background] Newman B, Selby JV, King MC, Slemenda C, Fabsitz R, Friedman GD. Concordance for type 2 (non-insulin-dependent) diabetes mellitus in male twins. Diabetologia. 1987 Oct;30(10):763-8. doi: 10.1007/BF00275741. PMID 3428496
- [Background] O'Rahilly SP, Nugent Z, Rudenski AS, Hosker JP, Burnett MA, Darling P, Turner RC. Beta-cell dysfunction, rather than insulin insensitivity, is the primary defect in familial type 2 diabetes. Lancet. 1986 Aug 16;2(8503):360-4. doi: 10.1016/s0140-6736(86)90052-8. PMID 2874367
- [Background] Taylor SI, Accili D, Imai Y. Insulin resistance or insulin deficiency. Which is the primary cause of NIDDM? Diabetes. 1994 Jun;43(6):735-40. doi: 10.2337/diab.43.6.735. No abstract available. PMID 8194657
- [Background] DeFronzo RA, Tobin JD, Andres R. Glucose clamp technique: a method for quantifying insulin secretion and resistance. Am J Physiol. 1979 Sep;237(3):E214-23. doi: 10.1152/ajpendo.1979.237.3.E214. PMID 382871
- [Background] Matthews DR, Hosker JP, Rudenski AS, Naylor BA, Treacher DF, Turner RC. Homeostasis model assessment: insulin resistance and beta-cell function from fasting plasma glucose and insulin concentrations in man. Diabetologia. 1985 Jul;28(7):412-9. doi: 10.1007/BF00280883. PMID 3899825
- [Background] Rizza RA, Mandarino LJ, Gerich JE. Mechanism and significance of insulin resistance in non-insulin-dependent diabetes mellitus. Diabetes. 1981 Dec;30(12):990-5. doi: 10.2337/diab.30.12.990. PMID 7030834
- [Background] Sherwin RS, Hendler RG, Felig P. Effect of diabetes mellitus and insulin on the turnover and metabolic response to ketones in man. Diabetes. 1976 Sep;25(9):776-84. doi: 10.2337/diab.25.9.776. PMID 955305
- [Background] DeFronzo RA, Ferrannini E. Insulin resistance. A multifaceted syndrome responsible for NIDDM, obesity, hypertension, dyslipidemia, and atherosclerotic cardiovascular disease. Diabetes Care. 1991 Mar;14(3):173-94. doi: 10.2337/diacare.14.3.173. PMID 2044434
- [Background] Luzi L, DeFronzo RA. Effect of loss of first-phase insulin secretion on hepatic glucose production and tissue glucose disposal in humans. Am J Physiol. 1989 Aug;257(2 Pt 1):E241-6. doi: 10.1152/ajpendo.1989.257.2.E241. PMID 2669517
- [Background] O'Rahilly S, Hattersley A, Vaag A, Gray H. Insulin resistance as the major cause of impaired glucose tolerance: a self-fulfilling prophesy? Lancet. 1994 Aug 27;344(8922):585-9. doi: 10.1016/s0140-6736(94)91969-0. PMID 7914964
- [Background] Lang DA, Matthews DR, Burnett M, Turner RC. Brief, irregular oscillations of basal plasma insulin and glucose concentrations in diabetic man. Diabetes. 1981 May;30(5):435-9. doi: 10.2337/diab.30.5.435. PMID 7014311
- [Background] Polonsky KS, Given BD, Hirsch LJ, Tillil H, Shapiro ET, Beebe C, Frank BH, Galloway JA, Van Cauter E. Abnormal patterns of insulin secretion in non-insulin-dependent diabetes mellitus. N Engl J Med. 1988 May 12;318(19):1231-9. doi: 10.1056/NEJM198805123181903. PMID 3283554
- [Background] Olefsky JM. Insulin resistance. In: Rifkin H, porte D Jr, eds. Ellenberg and Rifkin's diabetes mellitus: theory and practice. NewYork: Elsvier 1997: 513-52.
- [Background] Kolterman OG, Gray RS, Shapiro G, Scarlett JA, Griffin J, Olefsky JM. The acute and chronic effects of sulfonylurea therapy in type II diabetic subjects. Diabetes. 1984 Apr;33(4):346-54. doi: 10.2337/diab.33.4.346. PMID 6423429
- [Background] Lillioja S, Mott DM, Zawadzki JK, Young AA, Abbott WG, Knowler WC, Bennett PH, Moll P, Bogardus C. In vivo insulin action is familial characteristic in nondiabetic Pima Indians. Diabetes. 1987 Nov;36(11):1329-35. doi: 10.2337/diab.36.11.1329. PMID 3311855
- [Background] Garvey WT, Olefsky JM, Griffin J, Hamman RF, Kolterman OG. The effect of insulin treatment on insulin secretion and insulin action in type II diabetes mellitus. Diabetes. 1985 Mar;34(3):222-34. doi: 10.2337/diab.34.3.222. PMID 3882489
- [Background] Katsilambros N, Tentolouris N. Type 2 diabetes: an overview. In: Textbook of Diabetes, 3rd ed. Pickup JC and Williams G, Eds, Blackwell Science; 2003: pp 4.1-4.19.
- [Background] Gerich JE, Smith TM. beta-cell defects and pancreatic abnormalities in type 2 diabetes. In: Textbook of Diabetes, 3rd ed, Pickup JC & Williams G, Eds, Blackwell Science 23; 2003: 1-23.11.
- [Background] Armour T, Norris S, Brown D, Zhang X, Caspersen C. Initiating and maintaining physical activity for type 2 diabetes mellitus. Cochrane Database of Systematic Reviews 2004.
- [Background] Gimenez-Perez G, Gonzalez-Clemente JM, Mauricio D. Lifestyle interventions for preventing type 2 diabetes mellitus. Cochrane Database of Systematic Reviews 2001.
- [Background] Nield L, Summerbell CD, Hooper L, Whittaker V, Moore H. Dietary advice for the prevention of type 2 diabetes mellitus in adults. Cochrane Database Syst Rev. 2008 Jul 16;(3):CD005102. doi: 10.1002/14651858.CD005102.pub2. PMID 18646120
- [Background] Thomas DE, Elliott EJ, Naughton GA. Exercise for type 2 diabetes mellitus. Cochrane Database Syst Rev. 2006 Jul 19;2006(3):CD002968. doi: 10.1002/14651858.CD002968.pub2. PMID 16855995
- [Background] Black C, Donnelly P, McIntyre L, Royle PL, Shepherd JP, Thomas S. Meglitinide analogues for type 2 diabetes mellitus. Cochrane Database Syst Rev. 2007 Apr 18;2007(2):CD004654. doi: 10.1002/14651858.CD004654.pub2. PMID 17443551
- [Background] Saenz A, Fernandez-Esteban I, Mataix A, Ausejo M, Roque M, Moher D. Metformin monotherapy for type 2 diabetes mellitus. Cochrane Database Syst Rev. 2005 Jul 20;(3):CD002966. doi: 10.1002/14651858.CD002966.pub3. PMID 16034881
- [Background] Salpeter S, Greyber E, Pasternak G, Salpeter E. Risk of fatal and nonfatal lactic acidosis with metformin use in type 2 diabetes mellitus. Cochrane Database Syst Rev. 2003;(2):CD002967. doi: 10.1002/14651858.CD002967. PMID 12804446
- [Background] Meriden T. Progress with thiazolidinediones in the management of type 2 diabetes mellitus. Clin Ther. 2004 Feb;26(2):177-90. doi: 10.1016/s0149-2918(04)90017-3. PMID 15038941
- [Background] Misso ML, Egberts KJ, Page M, O'Connor D, Shaw J. Continuous subcutaneous insulin infusion (CSII) versus multiple insulin injections for type 1 diabetes mellitus. Cochrane Database Syst Rev. 2010 Jan 20;2010(1):CD005103. doi: 10.1002/14651858.CD005103.pub2. PMID 20091571
- [Background] Richter B, Neises G. 'Human' insulin versus animal insulin in people with diabetes mellitus. Cochrane Database Syst Rev. 2005 Jan 25;2005(1):CD003816. doi: 10.1002/14651858.CD003816.pub2. PMID 15674916
- [Background] Roberts D, Van NW, Chang H, Pohula W, MCheang, Moffatt M, et al. Glargine versus other basal insulins (NPH, Lente, or Ultralente) for the treatment of type 1 diabetes mellitus. Cochrane Database of Systematic Reviews 2005.
- [Background] Charlotte E, Mathis G. Inhaled insulin. Diabetes Health Center 2007, http://diabetes. webmd.com/inhaledinsulin.
- [Background] Dunn C, Curran MP. Inhaled human insulin (Exubera): a review of its use in adult patients with diabetes mellitus. Drugs. 2006;66(7):1013-32. doi: 10.2165/00003495-200666070-00019. PMID 16740022
- [Background] Smith U. Pioglitazone: mechanism of action. Int J Clin Pract Suppl. 2001 Sep;(121):13-8. PMID 11594239
- [Background] Yki-Jarvinen H. Thiazolidinediones. N Engl J Med. 2004 Sep 9;351(11):1106-18. doi: 10.1056/NEJMra041001. No abstract available. PMID 15356308
- [Background] Seda O, Sedova L. PPARs: molecular targets in the pharmacogenomics era. Prague Med Rep. 2004;105(3):223-36. PMID 15782550
- [Background] Kim H, Haluzik M, Asghar Z, Yau D, Joseph JW, Fernandez AM, Reitman ML, Yakar S, Stannard B, Heron-Milhavet L, Wheeler MB, LeRoith D. Peroxisome proliferator-activated receptor-alpha agonist treatment in a transgenic model of type 2 diabetes reverses the lipotoxic state and improves glucose homeostasis. Diabetes. 2003 Jul;52(7):1770-8. doi: 10.2337/diabetes.52.7.1770. PMID 12829645
- [Background] Tonelli J, Li W, Kishore P, Pajvani UB, Kwon E, Weaver C, Scherer PE, Hawkins M. Mechanisms of early insulin-sensitizing effects of thiazolidinediones in type 2 diabetes. Diabetes. 2004 Jun;53(6):1621-9. doi: 10.2337/diabetes.53.6.1621. PMID 15161771
- [Background] Ferre P. The biology of peroxisome proliferator-activated receptors: relationship with lipid metabolism and insulin sensitivity. Diabetes. 2004 Feb;53 Suppl 1:S43-50. doi: 10.2337/diabetes.53.2007.s43. PMID 14749265
- [Background] Mayerson AB, Hundal RS, Dufour S, Lebon V, Befroy D, Cline GW, Enocksson S, Inzucchi SE, Shulman GI, Petersen KF. The effects of rosiglitazone on insulin sensitivity, lipolysis, and hepatic and skeletal muscle triglyceride content in patients with type 2 diabetes. Diabetes. 2002 Mar;51(3):797-802. doi: 10.2337/diabetes.51.3.797. PMID 11872682
- [Background] Miyazaki Y, Mahankali A, Matsuda M, Mahankali S, Hardies J, Cusi K, Mandarino LJ, DeFronzo RA. Effect of pioglitazone on abdominal fat distribution and insulin sensitivity in type 2 diabetic patients. J Clin Endocrinol Metab. 2002 Jun;87(6):2784-91. doi: 10.1210/jcem.87.6.8567. PMID 12050251
- [Background] Hundal RS, Krssak M, Dufour S, Laurent D, Lebon V, Chandramouli V, Inzucchi SE, Schumann WC, Petersen KF, Landau BR, Shulman GI. Mechanism by which metformin reduces glucose production in type 2 diabetes. Diabetes. 2000 Dec;49(12):2063-9. doi: 10.2337/diabetes.49.12.2063. PMID 11118008
- [Background] Metformin. http://en.wikipedia.org/wiki/Metformin (accessed on 20 October 2011)
- [Background] Hamman RF. Genetic and environmental determinants of non-insulin-dependent diabetes mellitus (NIDDM). Diabetes Metab Rev. 1992 Dec;8(4):287-338. doi: 10.1002/dmr.5610080402. No abstract available. PMID 1307522
- [Background] Avogaro A. Insulin resistance: trigger or concomitant factor in the metabolic syndrome. Panminerva Med. 2006 Mar;48(1):3-12. PMID 16633326
- [Background] Parikh H, Groop L. Candidate genes for type 2 diabetes. Rev Endocr Metab Disord. 2004 May;5(2):151-76. doi: 10.1023/B:REMD.0000021437.46773.26. No abstract available. PMID 15041791
- [Background] Lohmueller KE, Pearce CL, Pike M, Lander ES, Hirschhorn JN. Meta-analysis of genetic association studies supports a contribution of common variants to susceptibility to common disease. Nat Genet. 2003 Feb;33(2):177-82. doi: 10.1038/ng1071. Epub 2003 Jan 13. PMID 12524541
- [Background] Stumvoll M, Goldstein BJ, van Haeften TW. Type 2 diabetes: principles of pathogenesis and therapy. Lancet. 2005 Apr 9-15;365(9467):1333-46. doi: 10.1016/S0140-6736(05)61032-X. PMID 15823385
- [Background] Staels B, Fruchart JC. Therapeutic roles of peroxisome proliferator-activated receptor agonists. Diabetes. 2005 Aug;54(8):2460-70. doi: 10.2337/diabetes.54.8.2460. PMID 16046315
- [Background] Spiegelman BM. PPAR-gamma: adipogenic regulator and thiazolidinedione receptor. Diabetes. 1998 Apr;47(4):507-14. doi: 10.2337/diabetes.47.4.507. PMID 9568680
- [Background] Dubuquoy L, Dharancy S, Nutten S, Pettersson S, Auwerx J, Desreumaux P. Role of peroxisome proliferator-activated receptor gamma and retinoid X receptor heterodimer in hepatogastroenterological diseases. Lancet. 2002 Nov 2;360(9343):1410-8. doi: 10.1016/S0140-6736(02)11395-X. PMID 12424006
- [Background] Olefsky JM. Treatment of insulin resistance with peroxisome proliferator-activated receptor gamma agonists. J Clin Invest. 2000 Aug;106(4):467-72. doi: 10.1172/JCI10843. No abstract available. PMID 10953021
- [Background] Fajas L, Auboeuf D, Raspe E, Schoonjans K, Lefebvre AM, Saladin R, Najib J, Laville M, Fruchart JC, Deeb S, Vidal-Puig A, Flier J, Briggs MR, Staels B, Vidal H, Auwerx J. The organization, promoter analysis, and expression of the human PPARgamma gene. J Biol Chem. 1997 Jul 25;272(30):18779-89. doi: 10.1074/jbc.272.30.18779. PMID 9228052
- [Background] Auwerx J. PPARgamma, the ultimate thrifty gene. Diabetologia. 1999 Sep;42(9):1033-49. doi: 10.1007/s001250051268. PMID 10447513
- [Background] Gouda HN, Sagoo GS, Harding AH, Yates J, Sandhu MS, Higgins JP. The association between the peroxisome proliferator-activated receptor-gamma2 (PPARG2) Pro12Ala gene variant and type 2 diabetes mellitus: a HuGE review and meta-analysis. Am J Epidemiol. 2010 Mar 15;171(6):645-55. doi: 10.1093/aje/kwp450. Epub 2010 Feb 23. PMID 20179158
- [Background] Stumvoll M, Haring H. The peroxisome proliferator-activated receptor-gamma2 Pro12Ala polymorphism. Diabetes. 2002 Aug;51(8):2341-7. doi: 10.2337/diabetes.51.8.2341. PMID 12145143
- [Background] Altshuler D, Hirschhorn JN, Klannemark M, Lindgren CM, Vohl MC, Nemesh J, Lane CR, Schaffner SF, Bolk S, Brewer C, Tuomi T, Gaudet D, Hudson TJ, Daly M, Groop L, Lander ES. The common PPARgamma Pro12Ala polymorphism is associated with decreased risk of type 2 diabetes. Nat Genet. 2000 Sep;26(1):76-80. doi: 10.1038/79216. PMID 10973253
- [Background] Deeb SS, Fajas L, Nemoto M, Pihlajamaki J, Mykkanen L, Kuusisto J, Laakso M, Fujimoto W, Auwerx J. A Pro12Ala substitution in PPARgamma2 associated with decreased receptor activity, lower body mass index and improved insulin sensitivity. Nat Genet. 1998 Nov;20(3):284-7. doi: 10.1038/3099. PMID 9806549
- [Background] Paracchini V, Pedotti P, Taioli E. Genetics of leptin and obesity: a HuGE review. Am J Epidemiol. 2005 Jul 15;162(2):101-14. doi: 10.1093/aje/kwi174. Epub 2005 Jun 22. PMID 15972940
- [Background] Vigouroux C, Fajas L, Khallouf E, Meier M, Gyapay G, Lascols O, Auwerx J, Weissenbach J, Capeau J, Magre J. Human peroxisome proliferator-activated receptor-gamma2: genetic mapping, identification of a variant in the coding sequence, and exclusion as the gene responsible for lipoatrophic diabetes. Diabetes. 1998 Mar;47(3):490-2. doi: 10.2337/diabetes.47.3.490. No abstract available. PMID 9519760
- [Background] Mori H, Ikegami H, Kawaguchi Y, Seino S, Yokoi N, Takeda J, Inoue I, Seino Y, Yasuda K, Hanafusa T, Yamagata K, Awata T, Kadowaki T, Hara K, Yamada N, Gotoda T, Iwasaki N, Iwamoto Y, Sanke T, Nanjo K, Oka Y, Matsutani A, Maeda E, Kasuga M. The Pro12 -->Ala substitution in PPAR-gamma is associated with resistance to development of diabetes in the general population: possible involvement in impairment of insulin secretion in individuals with type 2 diabetes. Diabetes. 2001 Apr;50(4):891-4. doi: 10.2337/diabetes.50.4.891. PMID 11289058
- [Background] Ek J, Andersen G, Urhammer SA, Hansen L, Carstensen B, Borch-Johnsen K, Drivsholm T, Berglund L, Hansen T, Lithell H, Pedersen O. Studies of the Pro12Ala polymorphism of the peroxisome proliferator-activated receptor-gamma2 (PPAR-gamma2) gene in relation to insulin sensitivity among glucose tolerant caucasians. Diabetologia. 2001 Sep;44(9):1170-6. doi: 10.1007/s001250100629. PMID 11596673
- [Background] Chuang LM, Hsiung CA, Chen YD, Ho LT, Sheu WH, Pei D, Nakatsuka CH, Cox D, Pratt RE, Lei HH, Tai TY. Sibling-based association study of the PPARgamma2 Pro12Ala polymorphism and metabolic variables in Chinese and Japanese hypertension families: a SAPPHIRe study. Stanford Asian-Pacific Program in Hypertension and Insulin Resistance. J Mol Med (Berl). 2001 Nov;79(11):656-64. doi: 10.1007/s001090100255. PMID 11715069
- [Background] Hara K, Yamauchi T, Kubota N, Tobe K, Yamazaki T, Nagai R, Kadowaki T. [The role of PPARgamma in the onset of type 2 diabetes]. Nihon Yakurigaku Zasshi. 2003 Oct;122(4):317-24. doi: 10.1254/fpj.122.317. Japanese. PMID 14501167
- [Background] Koch M, Rett K, Maerker E, Volk A, Haist K, Deninger M, Renn W, Haring HU. The PPARgamma2 amino acid polymorphism Pro 12 Ala is prevalent in offspring of Type II diabetic patients and is associated to increased insulin sensitivity in a subgroup of obese subjects. Diabetologia. 1999 Jun;42(6):758-62. doi: 10.1007/s001250051225. PMID 10382597
- [Background] Globerman H, Zauberman Y, Makarov T, Beamer BA, Yen CJ, Shuldiner AR, Harel C, Karnieli E. Analysis of the peroxisome proliferator activated receptor gamma (PPARgamma) gene in HAIRAN syndrome with obesity. Clin Endocrinol (Oxf). 2000 Apr;52(4):479-85. doi: 10.1046/j.1365-2265.2000.00950.x. PMID 10762291
- [Background] Masugi J, Tamori Y, Mori H, Koike T, Kasuga M. Inhibitory effect of a proline-to-alanine substitution at codon 12 of peroxisome proliferator-activated receptor-gamma 2 on thiazolidinedione-induced adipogenesis. Biochem Biophys Res Commun. 2000 Feb 5;268(1):178-82. doi: 10.1006/bbrc.2000.2096. PMID 10652233
- [Background] Werman A, Hollenberg A, Solanes G, Bjorbaek C, Vidal-Puig AJ, Flier JS. Ligand-independent activation domain in the N terminus of peroxisome proliferator-activated receptor gamma (PPARgamma). Differential activity of PPARgamma1 and -2 isoforms and influence of insulin. J Biol Chem. 1997 Aug 8;272(32):20230-5. doi: 10.1074/jbc.272.32.20230. PMID 9242701
- [Background] Stumvoll M, Wahl HG, Loblein K, Becker R, Machicao F, Jacob S, Haring H. Pro12Ala polymorphism in the peroxisome proliferator-activated receptor-gamma2 gene is associated with increased antilipolytic insulin sensitivity. Diabetes. 2001 Apr;50(4):876-81. doi: 10.2337/diabetes.50.4.876. PMID 11289055
- [Background] Boden G. Role of fatty acids in the pathogenesis of insulin resistance and NIDDM. Diabetes. 1997 Jan;46(1):3-10. PMID 8971073
- [Background] U.K. prospective diabetes study 16. Overview of 6 years' therapy of type II diabetes: a progressive disease. U.K. Prospective Diabetes Study Group. Diabetes. 1995 Nov;44(11):1249-58. PMID 7589820
- [Background] Brown JB, Conner C, Nichols GA. Secondary failure of metformin monotherapy in clinical practice. Diabetes Care. 2010 Mar;33(3):501-6. doi: 10.2337/dc09-1749. Epub 2009 Dec 29. PMID 20040656
- [Background] Holstein A, Seeringer A, Kovacs P. Therapy With Oral Antidiabetic Drugs: Applied pharmacogenetics. British Journal of Diabetes & Vascular Disease 2011;11:10. DOI: 10.1177/1474651410397583 (accessed on 20 October 2011).
- [Background] Cavaghan MK, Ehrmann DA, Byrne MM, Polonsky KS. Treatment with the oral antidiabetic agent troglitazone improves beta cell responses to glucose in subjects with impaired glucose tolerance. J Clin Invest. 1997 Aug 1;100(3):530-7. doi: 10.1172/JCI119562. PMID 9239399
- [Background] Kubo K. Effect of pioglitazone on blood proinsulin levels in patients with type 2 diabetes mellitus. Endocr J. 2002 Jun;49(3):323-8. doi: 10.1507/endocrj.49.323. PMID 12201216
- [Background] Li J, Tian H, Ren Y, et al. Effect of pioglitazone on first phase insulin secretion in type 2 diabetes mellitus and impaired glucose tolerance. Diabetes. 2003 (Abstract No 1212-P); 52 : A281.
- [Background] Diani AR, Sawada G, Wyse B, Murray FT, Khan M. Pioglitazone preserves pancreatic islet structure and insulin secretory function in three murine models of type 2 diabetes. Am J Physiol Endocrinol Metab. 2004 Jan;286(1):E116-22. doi: 10.1152/ajpendo.00331.2003. Epub 2003 Oct 7. PMID 14532171
- [Background] Al-Shali KZ, House AA, Hanley AJ, Khan HM, Harris SB, Zinman B, Mamakeesick M, Fenster A, Spence JD, Hegele RA. Genetic variation in PPARG encoding peroxisome proliferator-activated receptor gamma associated with carotid atherosclerosis. Stroke. 2004 Sep;35(9):2036-40. doi: 10.1161/01.STR.0000138784.68159.a5. Epub 2004 Jul 29. PMID 15284449
- [Background] Power AC. Diabetes mellitus.In: KasperDL, Fauci AS, Longo DL,Braunwald E, Hauser SL, Jameson JL (Eds). Harrison's Principles of Internal Medicine, 16th ed. McGraw-Hill; 2005: 2152-79.
- [Background] Kaku K. Efficacy and safety of therapy with metformin plus pioglitazone in the treatment of patients with type 2 diabetes: a double-blind, placebo-controlled, clinical trial. Curr Med Res Opin. 2009 May;25(5):1111-9. doi: 10.1185/03007990902820816. PMID 19309251
- [Background] Bailey CJ. Treating insulin resistance in type 2 diabetes with metformin and thiazolidinediones. Diabetes Obes Metab. 2005 Nov;7(6):675-91. doi: 10.1111/j.1463-1326.2005.00497.x. PMID 16219011
- [Background] Kahn SE, Haffner SM, Heise MA, Herman WH, Holman RR, Jones NP, Kravitz BG, Lachin JM, O'Neill MC, Zinman B, Viberti G; ADOPT Study Group. Glycemic durability of rosiglitazone, metformin, or glyburide monotherapy. N Engl J Med. 2006 Dec 7;355(23):2427-43. doi: 10.1056/NEJMoa066224. Epub 2006 Dec 4. PMID 17145742
- [Background] Schernthaner G, Matthews DR, Charbonnel B, Hanefeld M, Brunetti P; Quartet [corrected] Study Group. Efficacy and safety of pioglitazone versus metformin in patients with type 2 diabetes mellitus: a double-blind, randomized trial. J Clin Endocrinol Metab. 2004 Dec;89(12):6068-76. doi: 10.1210/jc.2003-030861. PMID 15579760
- [Background] Nagasaka S, Aiso Y, Yoshizawa K, Ishibashi S. Comparison of pioglitazone and metformin efficacy using homeostasis model assessment. Diabet Med. 2004 Feb;21(2):136-41. doi: 10.1111/j.1464-5491.2004.01083.x. PMID 14984448
- [Background] Tan MH, Glazer NB, Johns D, Widel M, Gilmore KJ. Pioglitazone as monotherapy or in combination with sulfonylurea or metformin enhances insulin sensitivity (HOMA-S or QUICKI) in patients with type 2 diabetes. Curr Med Res Opin. 2004 May;20(5):723-8. doi: 10.1185/030079904125003386. PMID 15140339
- [Background] Ceriello A, Johns D, Widel M, Eckland DJ, Gilmore KJ, Tan MH. Comparison of effect of pioglitazone with metformin or sulfonylurea (monotherapy and combination therapy) on postload glycemia and composite insulin sensitivity index during an oral glucose tolerance test in patients with type 2 diabetes. Diabetes Care. 2005 Feb;28(2):266-72. doi: 10.2337/diacare.28.2.266. PMID 15677777
- [Background] Yoon KH, Shin JA, Kwon HS, Lee SH, Min KW, Ahn YB, Yoo SJ, Ahn KJ, Park SW, Lee KW, Sung YA, Park TS, Kim MS, Kim YK, Nam MS, Kim HS, Park IeB, Park JS, Woo JT, Son HY. Comparison of the efficacy of glimepiride, metformin, and rosiglitazone monotherapy in korean drug-naive type 2 diabetic patients: the practical evidence of antidiabetic monotherapy study. Diabetes Metab J. 2011 Feb;35(1):26-33. doi: 10.4093/dmj.2011.35.1.26. Epub 2011 Feb 28. PMID 21537410
- [Background] Vilar L, Canadas V, Arruda MJ, Arahata C, Agra R, Pontes L, Montenegro L, Vilar CF, Silva LM, Albuquerque JL, Gusmao A. Comparison of metformin, gliclazide MR and rosiglitazone in monotherapy and in combination for type 2 diabetes. Arq Bras Endocrinol Metabol. 2010 Mar;54(3):311-8. doi: 10.1590/s0004-27302010000300010. PMID 20520962
- [Background] Ito H, Ohno Y, Yamauchi T, Kawabata Y, Ikegami H. Efficacy and safety of metformin for treatment of type 2 diabetes in elderly Japanese patients. Geriatr Gerontol Int. 2011 Jan;11(1):55-62. doi: 10.1111/j.1447-0594.2010.00635.x. PMID 20695906
- [Background] Kaku K, Tajima N, Kawamori R. Melbin observational research (MORE) study of metformin therapy in patients with type 2 diabetes mellitus. J Japan Diab Soc 2006; 49: 325-331 (in Japanese).
- [Background] Miyazaki Y, Matsuda M, DeFronzo RA. Dose-response effect of pioglitazone on insulin sensitivity and insulin secretion in type 2 diabetes. Diabetes Care. 2002 Mar;25(3):517-23. doi: 10.2337/diacare.25.3.517. PMID 11874940
- [Background] Matthews DR, Charbonnel BH, Hanefeld M, Brunetti P, Schernthaner G. Long-term therapy with addition of pioglitazone to metformin compared with the addition of gliclazide to metformin in patients with type 2 diabetes: a randomized, comparative study. Diabetes Metab Res Rev. 2005 Mar-Apr;21(2):167-74. doi: 10.1002/dmrr.478. PMID 15386821
- [Background] de Winter W, DeJongh J, Post T, Ploeger B, Urquhart R, Moules I, Eckland D, Danhof M. A mechanism-based disease progression model for comparison of long-term effects of pioglitazone, metformin and gliclazide on disease processes underlying Type 2 Diabetes Mellitus. J Pharmacokinet Pharmacodyn. 2006 Jun;33(3):313-43. doi: 10.1007/s10928-006-9008-2. Epub 2006 Mar 22. PMID 16552630
- [Background] Rasouli N, Raue U, Miles LM, Lu T, Di Gregorio GB, Elbein SC, Kern PA. Pioglitazone improves insulin sensitivity through reduction in muscle lipid and redistribution of lipid into adipose tissue. Am J Physiol Endocrinol Metab. 2005 May;288(5):E930-4. doi: 10.1152/ajpendo.00522.2004. Epub 2005 Jan 4. PMID 15632102
- [Background] Summerson JH, Bell RA, Konen JC. Coronary heart disease risk factors in black and white patients with non-insulin-dependent diabetes mellitus. Ethn Health. 1996 Mar;1(1):9-20. doi: 10.1080/13557858.1996.9961766. PMID 9395544
- [Background] Langenfeld MR, Forst T, Hohberg C, Kann P, Lubben G, Konrad T, Fullert SD, Sachara C, Pfutzner A. Pioglitazone decreases carotid intima-media thickness independently of glycemic control in patients with type 2 diabetes mellitus: results from a controlled randomized study. Circulation. 2005 May 17;111(19):2525-31. doi: 10.1161/01.CIR.0000165072.01672.21. Epub 2005 May 9. PMID 15883215
- [Background] Greene ME, Blumberg B, McBride OW, Yi HF, Kronquist K, Kwan K, Hsieh L, Greene G, Nimer SD. Isolation of the human peroxisome proliferator activated receptor gamma cDNA: expression in hematopoietic cells and chromosomal mapping. Gene Expr. 1995;4(4-5):281-99. PMID 7787419
- [Background] Elbrecht A, Chen Y, Cullinan CA, Hayes N, Leibowitz Md, Moller DE, Berger J. Molecular cloning, expression and characterization of human peroxisome proliferator activated receptors gamma 1 and gamma 2. Biochem Biophys Res Commun. 1996 Jul 16;224(2):431-7. doi: 10.1006/bbrc.1996.1044. PMID 8702406
- [Background] Matthaei S, Stumvoll M, Kellerer M, Haring HU. Pathophysiology and pharmacological treatment of insulin resistance. Endocr Rev. 2000 Dec;21(6):585-618. doi: 10.1210/edrv.21.6.0413. PMID 11133066
- [Background] Perriello G, Misericordia P, Volpi E, Santucci A, Santucci C, Ferrannini E, Ventura MM, Santeusanio F, Brunetti P, Bolli GB. Acute antihyperglycemic mechanisms of metformin in NIDDM. Evidence for suppression of lipid oxidation and hepatic glucose production. Diabetes. 1994 Jul;43(7):920-8. doi: 10.2337/diab.43.7.920. PMID 8013758
- [Background] Zhou G, Myers R, Li Y, Chen Y, Shen X, Fenyk-Melody J, Wu M, Ventre J, Doebber T, Fujii N, Musi N, Hirshman MF, Goodyear LJ, Moller DE. Role of AMP-activated protein kinase in mechanism of metformin action. J Clin Invest. 2001 Oct;108(8):1167-74. doi: 10.1172/JCI13505. PMID 11602624
- [Background] Moser M, Sowers JR. Clinical Management of Cardiovascular Risk Factors in Diabetes. 4th ed. USA: Professional Communications Publishing; 2011 : p 230.
- [Background] Nissen SE, Nicholls SJ, Wolski K, Nesto R, Kupfer S, Perez A, Jure H, De Larochelliere R, Staniloae CS, Mavromatis K, Saw J, Hu B, Lincoff AM, Tuzcu EM; PERISCOPE Investigators. Comparison of pioglitazone vs glimepiride on progression of coronary atherosclerosis in patients with type 2 diabetes: the PERISCOPE randomized controlled trial. JAMA. 2008 Apr 2;299(13):1561-73. doi: 10.1001/jama.299.13.1561. Epub 2008 Mar 31. PMID 18378631
- [Background] Wulffele MG, Kooy A, de Zeeuw D, Stehouwer CD, Gansevoort RT. The effect of metformin on blood pressure, plasma cholesterol and triglycerides in type 2 diabetes mellitus: a systematic review. J Intern Med. 2004 Jul;256(1):1-14. doi: 10.1111/j.1365-2796.2004.01328.x. PMID 15189360
- [Background] Seidell JC, Hautvast JG, Deurenberg P. Overweight: fat distribution and health risks. Epidemiological observations. A review. Infusionstherapie. 1989 Dec;16(6):276-81. doi: 10.1159/000222401. PMID 2696728
- [Background] O'Moore-Sullivan TM, Prins JB. Thiazolidinediones and type 2 diabetes: new drugs for an old disease. Med J Aust. 2002 Apr 15;176(8):381-6. doi: 10.5694/j.1326-5377.2002.tb04461.x. PMID 12041635
- [Background] Shihara N, Kitaoka M, Inagaki N, Kadowaki T, Koumoto S, Satoh J, Terauchi Y, Nunoi K, Yamada Y, Sakamaki H, Seino Y. Randomized controlled trial of single-agent glimepiride and pioglitazone in Japanese patients with type 2 diabetes: A comparative study. J Diabetes Investig. 2011 Oct 7;2(5):391-8. doi: 10.1111/j.2040-1124.2011.00115.x. PMID 24843519
- [Background] Kang ES, Park SY, Kim HJ, Kim CS, Ahn CW, Cha BS, Lim SK, Nam CM, Lee HC. Effects of Pro12Ala polymorphism of peroxisome proliferator-activated receptor gamma2 gene on rosiglitazone response in type 2 diabetes. Clin Pharmacol Ther. 2005 Aug;78(2):202-8. doi: 10.1016/j.clpt.2005.04.013. PMID 16084854
- [Background] Beamer BA, Yen CJ, Andersen RE, Muller D, Elahi D, Cheskin LJ, Andres R, Roth J, Shuldiner AR. Association of the Pro12Ala variant in the peroxisome proliferator-activated receptor-gamma2 gene with obesity in two Caucasian populations. Diabetes. 1998 Nov;47(11):1806-8. doi: 10.2337/diabetes.47.11.1806. No abstract available. PMID 9792554
- [Background] Ek J, Urhammer SA, Sorensen TI, Andersen T, Auwerx J, Pedersen O. Homozygosity of the Pro12Ala variant of the peroxisome proliferation-activated receptor-gamma2 (PPAR-gamma2): divergent modulating effects on body mass index in obese and lean Caucasian men. Diabetologia. 1999 Jul;42(7):892-5. doi: 10.1007/s001250051243. PMID 10440134
- [Background] Nicklas BJ, van Rossum EF, Berman DM, Ryan AS, Dennis KE, Shuldiner AR. Genetic variation in the peroxisome proliferator-activated receptor-gamma2 gene (Pro12Ala) affects metabolic responses to weight loss and subsequent weight regain. Diabetes. 2001 Sep;50(9):2172-6. doi: 10.2337/diabetes.50.9.2172. PMID 11522688
- [Background] Iwata E, Matsuda H, Fukuda T, Fukuen S, Motomura T, Igarashi T, Yamamoto I, Azuma J. Mutations of the peroxisome proliferator-activated receptor gamma (PPAR gamma) gene in a Japanese population : the Pro12Ala mutation in PPAR gamma 2 is associated with lower concentrations of serum total and non-HDL cholesterol. Diabetologia. 2001 Oct;44(10):1354-5. doi: 10.1007/s001250100647. No abstract available. PMID 11692187
- [Background] Oh EY, Min KM, Chung JH, Min YK, Lee MS, Kim KW, Lee MK. Significance of Pro12Ala mutation in peroxisome proliferator-activated receptor-gamma2 in Korean diabetic and obese subjects. J Clin Endocrinol Metab. 2000 May;85(5):1801-4. doi: 10.1210/jcem.85.5.6499. PMID 10843155
- [Background] Snitker S, Watanabe RM, Ani I, Xiang AH, Marroquin A, Ochoa C, Goico J, Shuldiner AR, Buchanan TA; Troglitazone in Prevention of Diabetes (TRIPOD) study. Changes in insulin sensitivity in response to troglitazone do not differ between subjects with and without the common, functional Pro12Ala peroxisome proliferator-activated receptor-gamma2 gene variant: results from the Troglitazone in Prevention of Diabetes (TRIPOD) study. Diabetes Care. 2004 Jun;27(6):1365-8. doi: 10.2337/diacare.27.6.1365. PMID 15161789
- See also: Bangladesh Institute of Research & Rehabilitation in Diabetes, Endocrine and Metabolic Disorders (BIRDEM) — http://www.birdem-bd.org/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Location: Bangladesh Institute of Research and Rehabilitation in Diabetes, Endocrine and Metabolic Disorders (BIRDEM),Dhaka, Bangladesh and National Forensic DNA Profiling Laboratory, Dhaka Medical College, Dhaka.
  Recruitment of patients were started at November 2008 and ended at December 2010.
Pre-assignment Details: 130 Type 2 Diabetes Mellitus (T2DM) out door patients of BIRDEM were screened to participate in the study.80 patients signed consent form and 77 enrolled the trial.3 patients didn't participate due to unknown cause.The patients were directed to follow their routine diet chart as before.
Groups:
- Single Group Study With Two Drugs- Pioglitazone and Metformin: Group 001-Pioglitazone 30 mg tablet once daily Group 002-Metformin 850 mg tablet once daily
  The single group study with a wash out period of one month with metformin 850 mg tablet once daily.
  77 patients started with pioglitazone(7 drop out)and after one month wash out period 70 patients started with metformin (9 drop out).
  48 patients for the 1st 3 months of pioglitazone and 32 patients for the 2nd 3 months of metformin responded to the drugs respectively according to the response rate[The treatment target was set to reduce at least ≥10% FBG or ≥1% HbA1c in the patients considering as the responder group].
Period: 001 (Pioglitazone) -3 Months
Arm/Group | Single Group Study With Two Drugs- Pioglitazone and Metformin
Started | 77
Completed | 70 (dropped out 7 patients)
Not Completed | 7
Not completed — Protocol Violation | 1
Not completed — Withdrawal by Subject | 1
Not completed — Lost to Follow-up | 2
Not completed — Lack of Efficacy | 1
Not completed — biasedness about the double blind method | 2
Period: 002 (Metformin)-3 Months
Arm/Group | Single Group Study With Two Drugs- Pioglitazone and Metformin
Started | 70 (70 patients participated for trial of drug 002.)
Completed | 61 (61 patients completed the drug 002.9 patients dropped out.)
Not Completed | 9
Not completed — Lack of Efficacy | 1
Not completed — Lost to Follow-up | 2
Not completed — Protocol Violation | 2
Not completed — Adverse Event | 2
Not completed — Husbands of female patients refrained | 2

BASELINE CHARACTERISTICS:
Groups:
- Single Group Study With Two Interventions: This was double blind, single group and "within subjects" designed study with two interventions.We screened 130 patients, selected 77 subjects who received drug Code 001, then gone through one month wash out period, then received Code 002.For PPARγ genotyping blood samples were collected from patients. There were found two groups-Pro12Pro and Pro12Ala. Baseline evaluation included detailed medical history,socioeconomic status, physical examination, and laboratory investigations for biomedical variables,psychosocial factors according to Patient Health Questionnaire (PHQ-9) and WHO-5 questionnaires.We decoded blinded drug after analyzing the results and knew that pioglitazone (30 mg once daily) was coded as 001 and metformin (850 mg once daily) as code 002.
  For statistical analysis we compare Pio vs Met, Pro12Pro vs Pro12Ala, met responder vs non responder.
Arm/Group | Single Group Study With Two Interventions
Number analyzed (Participants) | 77
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 77
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 46 (6.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47
  Male | 30
Region of Enrollment [Number; unit: participants]
  Bangladesh | 77

OUTCOME MEASURES:

1. Secondary Outcome: Comparison of Changes in Lipid Profiles With Pioglitazone and Metformin
Description: Response rate was defined by ≥10% decrease of FSG or/and ≥1% decrease of HbA1c from the baseline values after 3 months treatment.48 responded to pioglitazone and 32 responded to metformin.
  Analysis 1:Total Cholesterol(TC) Analysis 2:Triglyceride(TG) Analysis 3:High Density Lipoprotein(HDL) Analysis 4:Low Density Lipoprotein(LDL)
Time Frame: 3 months for each drug
Population: After completion of both of the treatments, it is found in the 3rd month some patients didn't response according to the response rate and during result analysis the responded numbers (48 and 32)were considered only. That's why the number of participant in both the trials didn't match with number of participants analyzed.
Measure: Mean (Standard Deviation); unit: mg/dl
Groups:
- Pioglitazone (001 Group): Dose: Pioglitazone tablet 30 mg once daily for 3 months
- Metformin (002 Group): Dose: Metformin tablet 850 mg once daily for 3 months
Arm/Group | Pioglitazone (001 Group) | Metformin (002 Group)
Number analyzed (Participants) | 48 | 32
mg/dl
  Baseline TC | 182.0 (44) | 193.0 (48.0)
  3rd month TC | 178 (42) | 177.0 (38.0)
  Baseline TG | 183 (128) | 166.0 (89.0)
  3rd month TG | 195 (165) | 175.0 (108.0)
  Baseline HDL | 33 (10) | 34.4 (9.0)
  3rd month HDL | 33.2 (8) | 34.7 (7.0)
  Baseline LDL | 112.8 (105.5) | 125.6 (47.0)
  3rd month LDL | 105.5 (47) | 112.0 (34.0)
Statistical Analysis 1: Comparison: Pioglitazone (001 Group) vs Metformin (002 Group); TC; Test type: Superiority or Other; p < 0.161, ANOVA — Category: Univariate & Multivariate analysis. (ANOVA, Pair t tests, MLR, OR, Pearson Correlation); Mean Difference (Net) = -9.06, 95% CI [-88.0 to 118], Standard Deviation 39.47
Statistical Analysis 2: Comparison: Pioglitazone (001 Group) vs Metformin (002 Group); TG; Test type: Superiority or Other; p < 0.913, ANOVA — Category: Univariate & Multivariate analysis. (ANOVA, Pair t tests, MLR, OR, Pearson Correlation); Mean Difference (Net) = 10.66, 95% CI 2-sided [-397.0 to 976], Standard Deviation 143.22
Statistical Analysis 3: Comparison: Pioglitazone (001 Group) vs Metformin (002 Group); HDL; Test type: Superiority or Other; p < 0.322, ANOVA — Category: Univariate & Multivariate analysis. (ANOVA, Pair t tests, MLR, OR, Pearson Correlation); Mean Difference (Net) = -0.47, 95% CI 2-sided [-35.0 to 19.0], Standard Deviation 9.59
Statistical Analysis 4: Comparison: Pioglitazone (001 Group) vs Metformin (002 Group); LDL; Test type: Superiority or Other; p < 0.210, ANOVA — Category: Univariate & Multivariate analysis. (ANOVA, Pair t tests, MLR, OR, Pearson Correlation); Mean Difference (Net) = -10.62, 95% CI 2-sided [-113.8 to 76.2], Standard Deviation 32.05

2. Primary Outcome: Comparison of Changes in Fasting Serum Glucose (FSG)With Pioglitazone and Metformin
Description: Response rate was defined by ≥10% decrease of FSG or/and ≥1% decrease of HbA1c from the baseline values after 3 months treatment.48 responded to pioglitazone and 32 responded to metformin.
Time Frame: 3 months for each drug
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/l
Groups:
- Pioglitazone (001 Group): Dose: Pioglitazone tablet 30mg once daily for 3 months.
- Metformin ( 002 Group): Dose: Metformin tablet 850 mg once daily for 3 months
Arm/Group | Pioglitazone (001 Group) | Metformin ( 002 Group)
Number analyzed (Participants) | 48 | 32
mmol/l
  Baseline FSG | 6.9 (2.5) | 6.2 (1.6)
  3rd Month FSG | 5.4 (1.2) | 6.5 (2.6)
Statistical Analysis 1: Comparison: Pioglitazone (001 Group) vs Metformin ( 002 Group); Change from Baseline in FSG at 3rd month; Test type: Superiority or Other; p < 0.05, ANOVA — Category: Univariate & Multivariate analysis. (ANOVA, Pair t tests, Multiple Logistic Regression (MLR), OR, Pearson Correlation); Mean Difference (Net) = -0.74, 95% CI 2-sided [-7.9 to 8.0], Standard Deviation 2.41 — The group 001 was divided according to Pro12Pro and Pro12Ala groups.There was no Ala12Ala group.These two groups were compared also in accordance with all parameters (glycemic levels, insulin levels, lipid profiles, BMI)

3. Primary Outcome: Comparison of Changes in Glycosylated Hemoglobin (HbA1c)With Pioglitazone and Metformin
Description: as for outcome 2
Time Frame: 3 months for each drug
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Pioglitazone (001 Group) | Metformin ( 002 Group)
Number analyzed (Participants) | 48 | 32
percentage
  Baseline HbA1c | 7.3 (1.2) | 7.8 (2.0)
  3rd month HbA1c | 6.7 (1.1) | 7.0 (1.5)
Statistical Analysis 1: Comparison: Pioglitazone (001 Group) vs Metformin ( 002 Group); Test type: Superiority or Other; p > 0.05, ANOVA — Category: Univariate & Multivariate analysis. (ANOVA, Pair t tests, MLR, OR, Pearson Correlation); Mean Difference (Net) = -0.64, 95% CI 2-sided [-4.4 to 2.4], Standard Deviation 1.07

4. Primary Outcome: Comparison of Changes in Insulin Levels (HOMA IR,QUICKI) With Pioglitazone and Metformin
Description: Response rate was defined by ≥10% decrease of FSG or/and ≥1% decrease of HbA1c from the baseline values after 3 months treatment.48 responded to pioglitazone and 32 responded to metformin.
  Analysis 1: Homeostasis Model Assessment Insulin Resistance(HOMA IR) Analysis 2: Quantitative Insulin sensitivity Check Index(QUICKI)
Time Frame: 3 months for each drug
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale ( SI unit)
Arm/Group | Pioglitazone (001 Group) | Metformin ( 002 Group)
Number analyzed (Participants) | 48 | 32
Score on a scale ( SI unit)
  Baseline QUICKI | 0.52 (0.08) | 0.57 (0.12)
  3rd month QUICKI | 0.59 (0.12) | 0.54 (0.09)
  Baseline HOMA IR | 5.1 (3.6) | 3.7 (2.9)
  3rd month HOMA IR | 2.9 (1.9) | 4.3 (3.6)
Statistical Analysis 1: Comparison: Pioglitazone (001 Group) vs Metformin ( 002 Group); Test type: Superiority or Other; p < 0.001, ANOVA — Category: Univariate & Multivariate analysis. (ANOVA, Pair t tests, MLR, OR, Pearson Correlation); Mean Difference (Net) = 0.02, 95% CI 2-sided [-0.40 to 0.27], Standard Deviation 0.12
Statistical Analysis 2: Comparison: Pioglitazone (001 Group) vs Metformin ( 002 Group); HOMA IR; Test type: Superiority or Other; p < 0.004, ANOVA — Category: Univariate & Multivariate analysis. (ANOVA, Pair t tests, MLR, OR, Pearson Correlation); Mean Difference (Net) = -1.04, 95% CI 2-sided [-14.12 to 15.52], Standard Deviation 4.25

5. Primary Outcome: Comparison of Changes in HOMA Percent B and HOMA Percent S With Pioglitazone and Metformin
Description: Response rate was defined by ≥10% decrease of FSG or/and ≥1% decrease of HbA1c from the baseline values after 3 months treatment.48 responded to pioglitazone and 32 responded to metformin.
  Analysis 1: Homeostatic Model Assessment of Beta cell function(HOMA percent B) Analysis 2: Homeostatic Model Assessment of Insulin Sensitivity (Homa percent S)
Time Frame: 3 months for each drug
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Pioglitazone (001 Group) | Metformin ( 002 Group)
Number analyzed (Participants) | 48 | 32
percentage
  Baseline HOMA percent beta cells function | 118.9 (87.0) | 109.3 (61.0)
  3rd month HOMA percent beta cells function | 132.3 (66.0) | 116.0 (77.0)
  Baseline HOMA percent sensitivity | 51.1 (30.8) | 76.2 (52.0)
  3rd month HOMA percent sensitivity | 69.3 (31.0) | 67.2 (45.0)
Statistical Analysis 1: Comparison: Pioglitazone (001 Group) vs Metformin ( 002 Group); HOMA B; Test type: Superiority or Other; p < 0.808, ANOVA — Category: Univariate & Multivariate analysis. (ANOVA, Pair t tests, MLR, OR, Pearson Correlation); Mean Difference (Net) = 9.79, 95% CI 2-sided [-346.40 to 328.10], Standard Deviation 84.46
Statistical Analysis 2: Comparison: Pioglitazone (001 Group) vs Metformin ( 002 Group); HOMA S; Test type: Superiority or Other; p < 0.025, ANOVA — Category: Univariate & Multivariate analysis. (ANOVA, Pair t tests, MLR, OR, Pearson Correlation); Mean Difference (Net) = 7.53, 95% CI 2-sided [-148.70 to 180], Standard Deviation 54.00

6. Primary Outcome: Comparison of Changes in Fasting Serum Insulin (FSI)With Pioglitazone and Metformin
Description: as for outcome 2
Time Frame: 3 months for each drug
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: μU/ml
Arm/Group | Pioglitazone (001 Group) | Metformin ( 002 Group)
Number analyzed (Participants) | 48 | 32
μU/ml
  Baseline FSI | 16.2 (8.7) | 13.0 (8.8)
  3rd month FSI | 12.3 (7.5) | 13.9 (7.3)
Statistical Analysis 1: Comparison: Pioglitazone (001 Group) vs Metformin ( 002 Group); FSI; Test type: Superiority or Other; p < 0.039, ANOVA — Category: Univariate & Multivariate analysis. (ANOVA, Pair t tests, MLR, OR, Pearson Correlation); Mean Difference (Net) = -2.09, 95% CI 2-sided [-27.04 to 26.52], Standard Deviation 10.2

ADVERSE EVENTS:
Time Frame: 3 months for pioglitazone treatment and next 3 months for metformin treatment
Groups:
- Pioglitazone (001 Group): 77 patients received the drug pioglitazone (30mg/day) for 3 months. Adverse events were assessed non-systematically on patients' complain generally and also systematically in case of hypertension, weight gain, common depression [Patient Health Questionnaire (PHQ-9) method] and creatinine increase.
  No serious adverse event was found during pioglitazone trial.
  In case of other adverse event, one patient complained for peripheral edema which disappeared (without medicine) within 2 days at the 2nd month of the treatment, Four patients gained weight within 10% of their initial weight after 3 months of the treatment and two patients complained for abdominal discomfort in the 1st month and normal treatment with antacid was provided to them.
- Metformin (002 Group): After wash out period 70 patients started with metformin (850mg/day) for further 3 months. Adverse events were assessed non-systematically on patients' complain and also systematically in case of hypertension, weight gain, common depression (PHQ-9 method) and creatinine increase.
  On basis of systemic data review and patient complain one patient was found with hypertension and another one was with increased creatinine level at the end of the metformin treatment and these events were assumed as serious adverse events as they were at health risk and withdrawn from the trial for intervention by hospital physician though they didn't need for hospitalization.
  One patient complained for mild diarrhea in the first month of the metformin treatment, the patient needed necessary treatment according to doctor's advice for one day, Five patients complained for abdominal discomfort in the 1st month and antacid was provided. Six patients were assumed suffering from common depression.
Arm/Group | Pioglitazone (001 Group) | Metformin (002 Group)
Serious Adverse Events (participants affected / at risk) | 0/77 | 2/70
Other Adverse Events (participants affected / at risk) | 14/77 | 19/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pioglitazone (001 Group) (N=77) | Metformin (002 Group) (N=70)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) — Systemic review of the data and patient's complain had shown that the patient's health was at risk. The patient was withdrawn in the 3rd month from the trial and referred to the hospital physician for proper treatment.
Creatinine increase (Renal and urinary disorders) | 0 (0) | 1 (1) — Patient's data review had shown the increase level of creatinine and was withdrawn from the trial in the 3rd month and referred to the hospital physician as it was assumed that its health was at risk.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pioglitazone (001 Group) (N=77) | Metformin (002 Group) (N=70)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2)
Backpain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 2 (2)
Headache (Nervous system disorders) | 1 (1) | 2 (2)
Common Depression (Nervous system disorders) | 3 (3) | 6 (6)
Peripheral Edema (Vascular disorders) | 1 (1) | 0 (0)
Weight gain (General disorders) | 4 (4) | 0 (0)
Mild Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 2 (2) | 5 (5)

LIMITATIONS AND CAVEATS:
The sample size was relatively small for more detailed analysis, treatment period was also short and there was a possibility of confounding by the use of non-study medication.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No